CLINICAL TRIAL: NCT04952051
Title: Randomized Controlled Blind End Point Study of Enalapril Folic Acid Tablets Combined With Calcium Antagonist or Diuretic to Prevent Stroke in Patients With Type H Hypertension
Brief Title: Enalapril Folic Acid Tablets Combined With CCB or Diuretic to Prevent Stroke in Patients With Type H Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: National Clinical Research Center, Southern Medical University (Unknown); Ningbo Yinzhou Community Health Service Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-132
Record Dates: First submitted 2021-06-20; First posted 2021-07-07 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enalapril Folic Acid Tablets Combined With amlodipine (Experimental): Enalapril Folic Acid Tablets 10.8mg Combined With amlodipine 5 or 10mg
  Interventions: Drug: Enalapril Folic Acid Tablets Combined With amlodipine
- Enalapril Folic Acid Tablets Combined With hydrochlorothiazide (Active Comparator): Enalapril Folic Acid Tablets 10.8mg Combined With hydrochlorothiazide 12.5 or 25mg
  Interventions: Drug: Enalapril Folic Acid Tablets Combined With hydrochlorothiazide

INTERVENTIONS:
Drug: Enalapril Folic Acid Tablets Combined With amlodipine — Enalapril Folic Acid Tablets 10.8mg Combined With amlodipine 5 or 10mg
  Arms: Enalapril Folic Acid Tablets Combined With amlodipine
Drug: Enalapril Folic Acid Tablets Combined With hydrochlorothiazide — Enalapril Folic Acid Tablets 10.8mg Combined With hydrochlorothiazide 12.5 or 25mg
  Arms: Enalapril Folic Acid Tablets Combined With hydrochlorothiazide

SUMMARY:
Hypertension is a common condition that can cause serious events such as stroke, coronary heart disease and heart failure. Homocysteine (Hcy) is a substance in the body that is harmful to blood vessels. Hyperhomocysteinemia (plasma Hcy≥10 mol/L), which is associated with hypertension, significantly increases the risk of stroke. This type of high blood pressure is called type "H" hypertension. Enalapril folic acid tablet is an innovative drug developed independently in China and is the first choice for the treatment of H type hypertension. Patients with type H hypertension should be treated with enalapril folic acid tablets to reduce stroke.

However, some patients had poor blood pressure control after monotherapy. At this time, other antihypertensive drugs should be used in combination. Amlodipine and Hydrochlorothiazide are the most commonly used and the best combination.

The purpose of this study was to observe the difference in the efficacy of enalapril folic acid tablets in patients with uncontrolled blood pressure who were well tolerated and randomized to aminoclodipine or hydrochlorothiazide in reducing stroke and other cardiovascular and cerebrovascular events, and to explore the relationship between various alternative measures and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 1.40-75 years old (inclusive);
* 2. Patients who have been diagnosed with all types of essential hypertension (those who are currently taking antihypertensive drugs with normal blood pressure can still be admitted) or those whose blood pressure screening meets the inclusion criteria;
* 3. Plasma (or serum) Hcy 10 mol/L;
* 4. Enalapril folic acid tablet 10.8 mg/day alone is not up to standard;
* 5. In the case of women of reproductive age, agree to use a reliable method of contraception during the trial;
* 6. Participate voluntarily and sign the informed consent;

Exclusion Criteria:

* 1. Previous stroke with definite diagnosis;
* 2. Patients with previous well-diagnosed myocardial infarction;
* 3. The presence of well-diagnosed heart failure;
* 4. Postoperative revascularization;
* 5.DBP >=110 mmHg or SBP >=180 mmHg;
* 6. Confirmed secondary hypertension;
* 7. Severe physical and systemic disease, which is estimated to be unable to complete the follow-up;
* 8. People with known congenital or acquired organic heart disease;
* 9. People who have had obvious intolerable adverse reactions to ACEI drugs in the past;
* 10. Have contraindications to ACEI drugs (including renal failure) or are allergic to the drugs used in the study or other ingredients in the drugs;
* 11. According to the researchers, there are contraindications to the use of folic acid;
* 12. Pregnant and lactating women;
* 13. If there are other obvious laboratory tests, abnormal physical signs and clinical diseases, it is not suitable to participate in the study according to the researcher's judgment;
* 14. Unwilling to participate in the trial, unwilling or unable to change the existing medication regimen;
* 15. Long-term use of folic acid or health medicines containing folic acid;
* 16.Severe mental disorder, unable to express their will

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Stroke rate | Until 5 years

SECONDARY OUTCOMES:
Rate of combined end points of cardiovascular events | Until 5 years
  Including cardiogenic death, cerebrovascular death, non-fatal stroke, and myocardial infarction
Rate of all causes of death | Until 5 years
  Including all causes and unexplained deaths
Rate of first or recurrent ischemic stroke | Until 5 years
Rate of first or recurrent hemorrhagic stroke | Until 5 years
Rate of myocardial infarction | Until 5 years

OTHER OUTCOMES:
Rate of heart failure (hospitalization) | Until 5 years
Rate of coronary revascularization | Until 5 years
Rate of peripheral arterial revascularization | Until 5 years
Rate of malignant tumor | Until 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, Study Chair — Second Affiliated Hospital of Zhejiang University, School of Medicine
Locations (1):
- Second affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China